CLINICAL TRIAL: NCT06805162
Title: Effect of an Unsupervised Multi-domain Intervention on Injury Risk Reduction in Athletics: Protocol of a Randomized Controlled Trial
Brief Title: Effect of an Unsupervised Multi-domain Intervention on Injury Risk Reduction in Athletics (I-ReductAI).
Acronym: I-ReductAI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Saint Etienne School of Mine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24CH262
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-02

CONDITIONS: Injury
Keywords: NEURO MUSCULAR; Athletics; injury prevention
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific training (Experimental): there will be a multi-domain intervention: i) A series of 12 educational videos on injury prevention; ii) Neuro-muscular exercise-based injury prevention programmes; iii) Techniques against stress and anxiety through breathing and mindfulness practice; iv) Injury prognostic feedback using individual data and based on a machine learning model.
  Interventions: Other: Specific training
- Normal training (Active Comparator): Athletes who continue their normal training
  Interventions: Other: Normal training

INTERVENTIONS:
Other: Normal training — Athletes should continue their normal training
  Arms: Normal training
Other: Specific training — Athletes should consider i) watching the educational videos on injury prevention, ii) perform the neuro-muscular exercises, iii) practice the techniques against stress and anxiety, and iv) consider the injury prognostic feedback.
  Arms: Specific training

SUMMARY:
In athletics, injuries can affect athletes' participation in athletics, their performance and career, but also their health in physical, psychological and social aspects, in the short, medium and long term.

DETAILED DESCRIPTION:
This justifies the development and implementation of injury risk reduction strategies. These should be developed according to a holistic approach that considers the complex aetiology of injuries in sport. Although many different injury risk reduction strategies have been studied in sport, in general, each has been evaluated in isolation, including for example education, neuromuscular exercises, psychological techniques or individual injury risk assessment. The investigators therefore hypothesized that their combination could improve the overall effectiveness of an intervention aimed at reducing the risk of injuries in athletics.

ELIGIBILITY:
Inclusion Criteria:

* be licensed at the French Athletics Federation (FFA) for competition (sprints, hurdles, jumps, throws, combined events, and endurance disciplines), without any counter-indications for competitive athletics activity attested by the license at the FFA;
* have daily access to a digital device (smartphone, computer, tablet) with a network connection (public or private).

Exclusion Criteria:

* Any athlete deprived of liberty or subject to legal protection (guardianship, under curatorship, legal protection).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 643 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-07-21 (Estimated); Study Completion 2025-07-21 (Estimated)

PRIMARY OUTCOMES:
Time (day) until the first Injury-type Complaint related to athletics and resulting in Restricted Participation in athletics (ICRP) | Week 14
  Time in days during which athletes are free of ICRP, between an intervention group and a control group

SECONDARY OUTCOMES:
Number of ICRP per 1000 hours of athletics practice | Week 14
  The number of ICRP per 1000 hours of athletics practice during a summer athletics competition season (14 weeks)
Number of days with an ICRP per 1000 hours of athletics practice | Week 14
  Number of days with ICRP per 1000 hours of athletics practice) during a summer athletics competition season (14 weeks)
Percentage of athletes with at least one ICRP | Week 14
  The percentage of athletes with at least one ICRP during a summer athletics competition season (14 weeks)
The average percentage of athletes with at least one ICRP | Week 14
  The average percentage of athletes with at least one ICRP per week during a summer athletics competition season (14 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: PASCAL EDOUARD, MD-PHD, Principal Investigator — CENTRE HOSPITALIER DE SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire, Saint-Etienne, France